CLINICAL TRIAL: NCT05003700
Title: Hepatic Arterial Infusion Chemotherapy Plus Lenvatinib and Camrelizumab for Unresectable Hepatocellular Carcinoma：a Prospective, Single-arm，Phase II Trial.
Brief Title: Hepatic Arterial Infusion Combined With Lenvatinib and Camrelizumab for Unresectable Hepatocellular Carcinoma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Nanfang Hospital, Southern Medical University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NFEC-2020-130
Record Dates: First submitted 2021-08-01; First posted 2021-08-12 (Actual); Last update posted 2024-11-05 (Actual); Status verified 2024-11

CONDITIONS: Hepatocellular Carcinoma
MeSH Terms: conditions — Carcinoma, Hepatocellular | interventions — lenvatinib; camrelizumab

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- HAIC(RALOX) plus Lenvatinib and Camrelizumab (Experimental): Hepatic arterial infusion of oxaliplatin and raltitrexed every 3 weeks. Lenvatinib 8 mg once daily (QD) oral dosing. Camrelizumab 200mg intravenously every 3 weeks.
  Interventions: Procedure: Hepatic arterial infusion chemotherapy; Drug: Lenvatinib; Drug: Camrelizumab

INTERVENTIONS:
Procedure: Hepatic arterial infusion chemotherapy — administration of oxaliplatin and raltitrexed via the tumor feeding arteries every 3 weeks.
Drug: Lenvatinib — 8 mg once daily (QD) oral dosing.
  Other Names: Lenvima
Drug: Camrelizumab — 200mg intravenously every 3 weeks.

SUMMARY:
The purpose of this study is to evaluate the efficacy and safety of hepatic arterial infusion chemotherapy of oxaliplatin and raltitrexed plus lenvatinib and camrelizumab in patients with unresectable hepatocellular carcinoma (HCC).

DETAILED DESCRIPTION:
Hepatic arterial infusion chemotherapy (HAIC) of oxaliplatin and raltitrexed was effective and safe for hepatocellular carcinoma. Lenvatinib was non-inferior to sorafenib in overall survival in untreated advanced hepatocellular carcinoma, and programmed cell death protein-1 (PD-1) antibody was effective and tolerable in patients with advanced hepatocellular carcinoma. No study has evaluated HAIC of oxaliplatin and raltitrexed plus lenvatinib and camrelizumab. Thus, the investigators carried out this prospective, single-arm study to find out it.

ELIGIBILITY:
Inclusion Criteria:

1. The patient voluntarily joins the study and signs an informed consent;
2. Age ≥ 18 years old, ≤ 75 years old, both men and women;
3. Clinical or pathologically confirmed BCLC B(tumor numbers≥4) or C-stage hepatocellular carcinoma, no further first-line treatment;
4. At least one intrahepatic evaluable tumor existed, intrahepatic tumor is the primary tumor burden;
5. Child-Pugh score small or equal to 7 points (Child-Pugh A-B);
6. The maximum liver tumor diameter ≥7cm;
7. ECOG score: 0 to 1 (according to the ECOG score classification);
8. The expected survival is longer than 12 weeks;
9. The laboratory parameters meets the following requirements (no blood components and cell growth factors are allowed within 14 days before the first dose):

   Absolute neutrophil count ≥ 1.5 × 109 / L; Platelets ≥ 50 × 109 / L; Hemoglobin ≥ 80 g / L; serum albumin ≥ 28 g / L; Thyroid stimulating hormone (TSH) ≤ 1 × ULN (if abnormalities should be considered at the same time FT3, FT4 levels, patients with FT3 and FT4 levels in normal range can also be enrolled); bilirubin ≤ 1.5 × ULN (within 7 days prior to the first dose); ALT ≤ 3 x ULN and AST ≤ 3 x ULN (within 7 days prior to the first dose); AKP ≤ 2.5 × ULN; serum creatinine ≤ 1.5 × ULN;
10. For female that non-surgical sterilization or in childbearing age need to use a medically approved contraceptive (such as an intrauterine device, contraceptive or condom) during the study period and within 3 months after the end of the study treatment period; For female that non-surgical sterilization or in childbearing age must have a negative serum or urine HCG test within 72 hours prior to study enrollment; and must be non-lactating; for male patients whose partner in a childbearing age, effective methods of contraception should be given during the trial and at the end of Camrelizumab injection.

Exclusion Criteria:

1. The patient has any active auto-immune disease or a history of auto-immune disease;
2. Evidence of hepatic decompensation including ascites, gastrointestinal bleeding or hepatic encephalopathy;
3. The patient is using immunosuppressive agents or systemic hormonal therapy for immunosuppression purposes (dose > 10 mg/day of prednisone or other therapeutic hormones) and continues to be used within 2 weeks prior to enrollment;
4. Known central nervous system tumors including metastatic brain disease;
5. Known history of HIV;
6. History of organ allograft;
7. Known or suspected allergy to the investigational agents or any agent given in association with this trial;
8. Suffering from hypertension, and cannot be well controlled by antihypertensive drugs (systolic blood pressure ≥ 140mmHg or diastolic blood pressure ≥90 mmHg);
9. Evidence of bleeding diathesis;
10. Patients with clinically significant gastrointestinal bleeding within 3 months prior to study entry.
11. Events of arterial/venous thrombosis occurring within the first 6 months of enrollment, such as cerebrovascular accidents (including transient ischemic attacks, cerebral hemorrhage, cerebral infarction), deep vein thrombosis, and pulmonary embolism;
12. Suffering heart diseases with clinical symptoms or those not well controlled, such as: (1) heart failure in NYHA class 2 or higher; (2) unstable angina; (3) myocardial infarction occurred within 1 year; (4) clinically symptomatic supraventricular or ventricular arrhythmia requiring treatment or intervention; (5) Tc > 450ms (male); QTc > 470ms (female);
13. Urine routine indicates that urine protein ≥ ++ and 24-hour urine protein amount > 1.0g was confirmed;
14. The patient has active infection, unexplained fever (≥38.5 °C) within 3 days before administration, or baseline white blood cell count>15×109/L;
15. Patients with congenital or acquired immunodeficiency (such as HIV-infected patients);
16. HBV-DNA>2000 IU/ml (or 104 copies/ml); or HCV-RNA>103 copies/ml; or HBsAg+ and anti-HCV antibody positive patients;
17. The patient has had other malignant tumors in the past 3 years or at the same time (except for cured skin basal cell carcinoma and cervical carcinoma in situ);
18. Patients have previously received other anti-PD-1 antibody therapy or other immunotherapy against PD-1/PD-L1, or have received apatinib before;
19. Inoculation of a live vaccine within less than 4 weeks prior to study or possibly during the study period;
20. Pregnant or lactating women, or women of childbearing age who are unwilling to take contraceptive measures;
21. According to the investigators, the patient has other factors that may affect the results of the study or lead to the termination of the study, such as alcohol abuse, drug abuse, other serious diseases (including mental illness) requiring combined treatment, and serious laboratory tests, abnormalities, accompanied by factors such as family or society, which may affect the safety of enrolled patients.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 39 (Actual)
Dates: Start 2021-08-12 (Actual); Primary Completion 2023-05-26 (Actual); Study Completion 2024-07-04 (Actual)

PRIMARY OUTCOMES:
Objective response rate (ORR) | From date of first dose of study drug until disease progression, development of unacceptable toxicity, withdrawal of consent, or sponsor termination (up to approximately 3 years)
  ORR is defined as the percentage of participants who have best overall response (BOR) of complete response (CR) or partial response (PR) at the time of data cutoff as assessed by RECIST 1.1

SECONDARY OUTCOMES:
The disease control rate (DCR) | From date of first dose of study drug until disease progression, stable disease, development of unacceptable toxicity, withdrawal of consent, or sponsor termination (up to approximately 3 years)
  DCR is defined as the percentage of participants who have best overall response (BOR) of complete response (CR) or partial response (PR) or stable disease (SD) at the time of data cutoff as assessed by RECIST 1.1
Duration of response (DOR) | From the first documentation of CR or PR to the first date of documentation of disease progression or death whichever occurs first (up to approximately 3 years)
  DOR is defined as the time from the first documentation of CR or PR to the date of first documentation of disease progression or death (whichever occurs first) as assessed by RECIST 1.1
Progression free survival rate at 12 months | From date of first dose of study drug to the date of first documentation of disease progression or death, whichever occurs first (up to approximately 3 years)
  The progression free survival time defined as the time from the first study dose date to the date of first documentation of disease progression as assessed by RECIST 1.1
Overall survival rate at 12 months | From date of first dose of study drug to the date of first documentation of death from any cause, whichever occurs first (up to approximately 3 years)
  OS is measured from the start date of the Treatment Phase (date of first study dose) until date of death from any cause. Participants who are lost to follow-up and the participants who are alive at the date of data cutoff will be censored at the date the participant was last known alive or the cut-off date, whichever comes earlier.
The median progression free survival time (mPFS) | From date of first dose of study drug to the date of first documentation of disease progression (up to approximately 3 years)
  The progression free survival time (mPFS) defined as the time from the first study dose date to the date of first documentation of disease progression as assessed by RECIST 1.1
The median overall survival time (mOS) | From the start date of the Treatment Phase until date of death from any cause (up to approximately 3 years)
  OS is measured from the start date of the Treatment Phase (date of first study dose) until date of death from any cause. Participants who are lost to follow-up and the participants who are alive at the date of data cutoff will be censored at the date the participant was last known alive or the cut-off date, whichever comes earlier.
Number of participants with treatment-related adverse events as assessed by CTCAE v5.0 | From the start date of the Treatment Phase until date of death from any cause (up to approximately 3 years)
  Safety will be evaluated according to the NCI CTCAE Version 5.0. All observations pertinent to the safety of the study medication will be recorded on the CRF and included in the final report.

CONTACTS AND LOCATIONS:
Overall Officials: Jinzhang Chen, Study Director — Nanfang Hospital, Southern Medical University
Locations (1):
- Nanfang Hospital of Southern Medical University, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: No